CLINICAL TRIAL: NCT04489576
Title: Efficacy and Safety of Keratin Hair Therapy on the Health of Hair and Scalp
Brief Title: Evaluation of Safety and Efficacy of Keratin Hair Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Abdelhamed, Associate professor, Department of Dermatology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sohagu310
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Hair Damage
Keywords: Hair keratin; Hair straightening

STUDY DESIGN:
Intervention Model Description: Keratin hair application
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigator and the outcome assessor will be blinded as regards the outcome measures evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (1): Treatment with keratin cure hair (Active Comparator): Group (1): Patients will be treated with Keratin cure ® hair treatment. It will be applied once with use of a flat iron.
  Interventions: Procedure: Keratin hair treatment (Keratin Cure ®) versus (QOD Max ®)
- Group (2): Treatment with Qod max keratin hair (Active Comparator): Group (2): Patients will be treated with QOD Max ® keratin hair treatment. It will be applied once with use of a flat iron.
  Interventions: Procedure: Keratin hair treatment (Keratin Cure ®) versus (QOD Max ®)
- Group (3): Treatment without keratin hair treatment (Placebo Comparator): Group (3): Patients will be treated without keratin hair treatment, but the same steps of keratin application will be followed.
  Interventions: Procedure: Keratin hair treatment (Keratin Cure ®) versus (QOD Max ®)

INTERVENTIONS:
Procedure: Keratin hair treatment (Keratin Cure ®) versus (QOD Max ®) — Hair will be treated with 2 different types of keratin in groups 1 & 2. All steps of keratin application will be done in group 3 without keratin application as a control group.
  Other Names: Hair straightening treatment

SUMMARY:
Hair appearance is an important issue for females. Treatment of hair with keratin has been popular among females nowadays. Although chemical hair straightening application has a beneficial effect on hair shafts with the repair of the broken cuticle, some side effects may occur. Therefore, this study aims to study the efficacy and safety of such new non-formaldehyde widely used keratin treatments on hair by assessment of changes of the scalp, hair density, and the morphology, color, and ultrastructure of hair shaft after application.

DETAILED DESCRIPTION:
Hair is an important feature for most women that contribute to one's individual identity. The appearance and morphology of the hair is one of the divergent traits in humans. Keratin in hair care products has two effects; it can penetrate the cortex of the hair fiber improving the mechanical properties of damaged fibers and promotes a surface coating that prevents or decreases water diffusion through the hair fibers.These properties have beneficial effects on the hair structure replacing lost keratin.However, the side effects and safety of this treatment have not yet been completely evaluated.There are many different brands of the keratin hair treatment, all with nearly the same basic chemical composition. Non-formaldehyde containing keratin straightening products, also known as safe keratin treatments (SKT) have recently been introduced to the market.Therefore, this study aims to study the efficacy and safety of such new non formaldehyde widely used keratin treatments on hair.

ELIGIBILITY:
Inclusion Criteria:

* The study will include female patients aged between 18 and 55 years, with hair curl types from III to V according to L'Oréal Curl Classification. The Patients will be randomized by simple randomization into 3 groups, 10 patients for each.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients having hair loss or under treatment of hair loss in last 3 months.
* Patients with previous history of keratin treatment.
* Patients with scalp affection including infection, injury or surgery
* Patients with chronic medical diseases.
* Patients with anemia (hemoglobin level <10mg/dl) or under its treatment.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants will be included as females are more interested in keratin hair straightening.
Enrollment: 30 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change of hair shedding using the Visual analogue scale (VAS) | Baseline, 2 months, 4 months, 6 months
  It will be used to evaluate hair shedding. Hair shedding is scored on a scale of 1-6. Women are asked to look at the scale and point to the photograph that best correlates with the amount of hair shed on an average day. Grades 1-3 are considered normal. Grade 4 is borderline, while Grades 5 and 6 indicate excessive shedding.
Change of hair morphology using trichoscope | Baseline, 2 months, 4 months, 6 months
  It will be used to evaluate hair structure and scalp. Hair density/cm 2 and thickness (mm) will be measured in the frontal, temporal and vertex areas in all participants.
Change of hair morphology using Transmission Electron Microscopic examination | Baseline, 2 months, 4 months, 6 months
  Randomly selected samples of each group will be fixed in 3% glutaraldehyde for over a period of 4 hours at 4°C and processed to be examined by transmission electron microscope
Safety evaluation | at 6 months
  to detect any side effects that will be reported either by the patient or by the physician.

SECONDARY OUTCOMES:
Change of patient satisfaction questionnaire about keratin treatment | Baseline, 2 months, 4 months, 6 months
  A 5 items Questionnaire will be completed by the patients to evaluate their satisfaction about the treatment. The questionnaire consists of Q1 (1-5), Q2,3 (1-7), Q4 (1-4) and Q5 has 3 sub-items Q5a, Q5b, Q5c (1-5 for each). Total score ranges from 7-38. Higher scores are associated with higher dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abdelhamed, MD, Principal Investigator — Faculty of Medicine, Sohag University, Egypt
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data sharing plan will include the study protocol, statistical analysis plan, and the clinical study report.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6 months after finishing the study.